CLINICAL TRIAL: NCT01468311
Title: Phase I/II Trial of Yttrium-90-labeled Daclizumab (Anti-CD25) Radioimmunotherapy With High-dose BEAM Chemotherapy and Autologous Hematopoietic Stem Cell Rescue in Recurrent and Refractory Hodgkin's Lymphoma
Brief Title: Yttrium-90-labeled Daclizumab With Chemotherapy and Stem Cell Transplant for Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Poor enrollment and ability to radioconjugate Daclizumab. Neither Center for Cancer Research (CCR) or Nuclear Medicine/Radiology wanted to do the facilities upgrade and hire personnel needed to radioconjugate the drug at the Clinical Center.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kevin Conlon, MD, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120003; 12-C-0003
Record Dates: First submitted 2011-11-05; First posted 2011-11-09 (Estimated); Results first posted 2017-05-25 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Hodgkin Disease; Hodgkin Lymphoma
Keywords: Immunotherapy; Resistant Hodgkins Lymphoma; Auto Stem Cell Transplant; Combination Chemo and Radiolabeled Monoclonal Antibody; Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Yttrium-90-labeled Daclizumab + Chemotherapy (Experimental): Yttrium-90-labeled Daclizumab + BCNU, etoposide, cytarabine and melphalan (BEAM) + Auto stem cell transplant (ASCT)
  Interventions: Procedure: Auto stem cell transplant; Drug: BEAM; Radiation: 111In-daclizumab; Radiation: 90Y-daclizumab

INTERVENTIONS:
Procedure: Auto stem cell transplant — Auto stem cell transplant (ASCT) is given after 90Y-daclizumab
Drug: BEAM — BCNU, etoposide, cytarabine and melphalan (BEAM) chemotherapy are given after 90Y-daclizumab
Radiation: 111In-daclizumab — 111In-daclizumab will be administered to patients with each therapeutic infusion of 90Y-daclizumab in order to define the distribution of radiolabeled daclizumab, and to allow visualization by scans.
Radiation: 90Y-daclizumab — 90Y-daclizumab administered with a fixed dose of pentetate calcium trisodium (Ca-DTPA) followed by BEAM Chemo and Auto stem cell transplant

SUMMARY:
Background:

* Hodgkins lymphoma (HL) is a highly treatable cancer. However, if HL does not respond to chemotherapy or returns after chemotherapy, further treatments often are not successful.
* Some HL cells have a molecule called cluster of differentiation 25 (CD25) on the surface. Daclizumab is a drug that can detect CD25 on cells. In a treatment study for HL that did not respond to chemotherapy, daclizumab plus a radioactive atom called Yttrium 90 helped kill these HL cells. Researchers want to combine this 90Y daclizumab with high-dose chemotherapy and stem cell transplant. This treatment may be more effective than the daclizumab alone.

Objectives:

- To see if yttrium-90 daclizumab, high-dose chemotherapy, and stem cell transplants can treat HL that has not responded to earlier treatments.

Eligibility:

- Individuals at least 18 years of age who have Hodgkins lymphoma that has not responded to chemotherapy.

Design:

* Participants will be screened with a physical exam and medical history. They will also have blood and urine tests.
* Participants will have filgrastim and plerixafor to move stem cells into the blood. Stem cells will be collected with apheresis.
* Four weeks after stem cells are collected, participants will have the 90Y daclizumab and normal daclizumab to treat the HL. Chemotherapy will start 9 days after the first treatment.
* Most participants will have a second dose of 90Y daclizumab 6 weeks after the first dose.
* After each daclizumab treatment, participants will have several imaging studies of the chest and abdomen. Blood samples will also be collected.
* On the day after the last day of chemotherapy, participants will receive the stem cells collected earlier. Filgrastim injections will help stimulate stem cell growth....

DETAILED DESCRIPTION:
Background:

* Although Hodgkins lymphoma (HL) is considered a highly treatable cancer, patients with relapsed and chemotherapy refractory disease represent a major therapeutic challenge.
* Only 30-65% of relapsed patients will achieve long-term disease free survival with the current standard of care high-dose chemotherapy with autologous hematopoietic stem cell transplant (ASCT).
* The malignant Reed-Sternberg cells of HL and the surrounding benign T cell infiltrates often express CD25, the high affinity interleukin-2 receptor (IL-2R alpha).
* In study NCI-97-C-0110, we treated 30 patients with CD25-expressing relapsed or refractory HL with radioimmunotherapy (RIT) using (90)Y-labeled daclizumab (anti-CD25), and achieved a 63% response rate including 12 complete responses with few serious adverse events other than MDS in 4 patients.
* We propose integrating (90)Y-labeled daclizumab RIT into the induction regimen of ASCT in an effort to improve the response and disease-free survival in relapsed and refractory HL.

Objectives:

Phase I Primary Objectives:

* To assess the safety and adverse events associated with (90)Y-daclizumab (humanized anti-CD25) radioimmunotherapy (RIT) in combination with high-dose BEAM (carmustine, etoposide, cytarabine, [Ara-C, cytosine arabinoside] and melphalan) chemotherapy and autologous hematopoietic stem cell transplantation (ASCT) in patients with relapsed or refractory Hodgkin s lymphoma (HL) with adverse prognostic factors.
* To determine the maximum tolerated dose in mCi of (90)Y-daclizumab RIT in combination with high-dose BEAM chemotherapy and ASCT in patients with relapsed or refractory HL.

Phase II Primary Objectives:

* To assess the frequency of the failure to engraft, myelodysplastic syndrome (MDS), secondary leukemia for the development of abnormal bone-marrow cytogenetics in refractory or relapsed HL patients treated with (90)Y-daclizumab RIT in combination with high-dose BEAM chemotherapy and ASCT.
* To estimate the response rate (the number of complete and partial responses) in patients with refractory or relapsed HD to (90)Y-daclizumab RIT administered in combination with high-dose BEAM chemotherapy and ASCT.

Eligibility:

* Patients must have a confirmed diagnosis of relapsed or refractory HL with at least 10% of malignant Reed-Sternberg cells or infiltrating T-cells expressing CD25 (IL-2R alpha). A. Patients must have at least one of the following: (1) had an initial relapse less than 12 months after achieving a complete response (CR) with primary chemotherapy for HL; (2) were Staged at III/IV at diagnosis; (3) exhibited chemotherapy resistant disease or (4) did not achieve a CR with cytoreductive chemotherapy prior to a planned transplant. B. Patient must have a lesion of at least 1.0 cm in its greatest diameter. C. Patients with lymphocyte predominant HL are excluded. D. Patients with pre-existing myelodysplastic syndrome (MDS) or marrow cytogenic abnormalities will not be eligible to participate.
* Omission of cytotoxic chemotherapy or other systemic therapy of HL for at least 4 weeks prior to entry into the trial.
* No prior ASCT or allogeneic stem cell transplant.

Design:

* A single institution non-randomized open-label phase I/II trial.
* Patients will undergo peripheral blood stem cell (PBSC) mobilization with granulocyte-colony stimulating factor (G-CSF, filgrastim) and Plerixafor followed by apheresis to collect a target dose of 4 x 106 cluster of differentiation 34 (CD34) cells/kg (minimal dose of 2 x 106 CD34+ cells/kg) of actual body weight.
* Phase I study will be carried out using a standard 3 + 3 cohort dose-escalation design:

  * Dose level 1: Patients will receive a single dose of 15 mCi 90Y-daclizumab RIT (day -15 2 days) followed by high-dose BEAM chemotherapy (beginning Day -6) and ASCT (Day 0).
  * Dose levels 2-7: Patients will receive two doses of 90Y-daclizumab RIT 6 weeks apart (Day -56 and -15 2 days) followed by high-dose BEAM chemotherapy (beginning day -6) and ASCT (Day 0). The first dose of 90Y-daclizumab will be fixed at 15 mCi. The second dose will be escalated in 15 mCi increments from 15 mCi until maximum tolerated dose, not to exceed 90 mCi.
* Phase II: All patients will receive two doses of 90Y-daclizumab (Day -56 and -15 2 days) followed by high-dose BEAM chemotherapy (beginning Day -6) and ASCT (Day 0). The first dose of RIT will be 15 mCi. The second dose will be the maximum tolerated dose as determined from phase I.

  111In-daclizumab (5 mCi) imaging may be performed concurrently with each 90Ydaclizumab RIT and at day 100 after ASCT.

ELIGIBILITY:
* INCLUSION CRITERIA:

2.1.1.1 All patients must have a pathologically confirmed diagnosis of classical Hodgkin's lymphoma (HL) as outlined in the World Health Organization (WHO) Classification System of Lymphoid Tumours. Patients with nodular lymphocyte-predominant Hodgkin's lymphoma (HL) (NLPHL) are not eligible.

2.1.1.2 Refractory or relapsed HL patients that are also candidates for auto stem cell transplant (ASCT).

2.1.1.3 At least one adverse prognostic factor: (1) initial relapse less than or equal to 12 months after primary chemotherapy, (2) staged as Ann Arbor Classification initial stage III or IV disease, (3) chemotherapy resistant disease, (4) Failure to achieve a complete response (CR) with cytoreductive chemotherapy or persistent positive (18) fluorodeoxyglucose positron emission tomography (FDGPET) imaging.

2.1.1.4 At least 10% of the cells obtained from lymph node, or extranodal sites must react with anti-cluster of differentiation 25 (CD25) (anti-Tac) on immunofluorescent or immunoperoxidase staining. Because of the high frequency of CD25 positivity of the infiltrating Tcells in HL tumors, patients with CD25-positive infiltrating T cells will be eligible even if their Hodgkin's (Reed-Sternberg) cells are CD25-negative.

2.1.1.5 Measurable disease as defined by the Cheson Response Criteria for Malignant Lymphoma detailed in section 6.2 with at least one lesion greater than or equal to 1.0 cm in longest diameter by computed tomography (CT) scan.

2.1.1.6 Omission of cytotoxic chemotherapy or other systemic therapy of the malignancy for greater than or equal to 4 weeks prior to entry into the trial. Patients must be greater than or equal to 4 weeks since major surgery, radiotherapy, or biotherapy/targeted therapies and recovered from the toxicity of prior treatment to less than or equal to CTC grade 1, exclusive of grade 2 alopecia, fatigue, lymphopenia, cluster of differentiation 4 (CD4)+ circulating T cells, white blood cell (WBC) or bilirubin.

2.1.1.7 Patients must be greater than or equal to 18-years old.

2.1.1.8 Patients must have a life expectancy of greater than 3 months.

2.1.1.9 Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 1.

2.1.1.10 The patient must have a granulocyte count of at least 1,500/microL and a platelet count of greater than 100,000/microL.

2.1.1.11 Patients must have a creatinine of less than 2.0 mg/dL, or if the patient has a serum creatinine greater than or equal to 2.0, a measured creatinine clearance (Ccr) must be greater than 60 mL/min/1.73m(2).

2.1.1.12 Patients must have a serum alkaline phosphatase, alanine aminotransferase (ALT) serum glutamic oxaloacetic transaminase (SGOT), and aspartate aminotransferase (AST) serum glutamic pyruvic transaminase (SGPT) less than 3 times the upper limit of normal (ULN), unless due to liver or bone involvement by HL. Under these circumstances, serum alkaline phosphatase, SGPT and SGOT must be less than 5 times ULN.

2.1.1.13 Patients must have a total serum bilirubin less than 2.5 times ULN.

2.1.1.14 Patients must have a cardiac ejection fraction greater than 45% on 2D echocardiography or multi-gated acquisition scan (MUGA) obtained within 28 days of study enrollment.

2.1.1.15 Lung diffusion capacity for carbon monoxide (DLCO) greater than 50%, or forced expiratory volume at 1.0 seconds (FEV1.0) greater than 65% of predicted on pulmonary function testing (PFT) obtained within 28 days of study enrollment.

2.1.1.16 Women of childbearing potential must have a negative serum Beta-human chorionic gonadotropin (HCG) pregnancy test at initial screening and within 3 days prior to registration.

2.1.1.17 The effects of (90)Y-daclizumab on the developing human fetus are unknown. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, while receiving treatment and for 4 months after undergoing ASCT. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

2.1.1.18 Patients receiving a stable dose (greater than 4 weeks) of corticosteroid therapy equivalent to 20 mg of prednisone per day or less are eligible.

2.1.1.19 Patients must be able to understand and sign informed consent.

EXCLUSION CRITERIA:

2.1.2.1 Patients who have relapsed from their initial Adriamycin, bleomycin, vinblastine, dacarbazine) ABVD or similar standard treatment regimen and have not received any other chemotherapy or salvage systemic treatment.

2.1.2.2 Patients that have received prior radioimmunotherapy.

2.1.2.2. Patients enrolled on another therapeutic study.

2.1.2.3 Patients that have received prior radioimmunotherapy.

2.1.2.4 Patients that have received a prior autologous or allogeneic stem cell transplant

2.1.2.5.Patients that have received prior radiation to the lung, excluding prior mediastinal

radiation.

2.1.2.6 Patients with greater than 25% involvement of the bone marrow with HL.

2.1.2.7 Patients with evidence of myelodysplasia, leukemia by morphology, immunostains flow cytometry or abnormal cytogenetics on a bone- marrow aspirate or biopsy. The diagnosis of myelodysplasia will be made by an independent investigator of the Laboratory of Pathology, National Cancer Institute (NCI) taking into consideration the totality of the clinical, pathological, flow cytometric and cytogenetic information described in Appendix E and present in a particular individual s evaluation.

2.1.2.8 Patients with history of central nervous system (CNS) involvement or active CNS involvement by malignancy.

2.1.2.9 Patients with an active second primary cancer will not be eligible. Patients curatively treated for a second cancer greater than 5 years prior to enrollment without a recurrence are eligible. Patients curatively treated for a second primary cancer within the last 5 years with a less than or equal to 5% risk of recurrence are eligible. Patients with a history of curatively treated basal cell carcinoma or intraepithelial neoplasia of the uterine cervix will be allowed on study.

2.1.2.10 Patients with serum human anti-human antibody (HAHA) against daclizumab.

2.1.2.11 Patients with human immunodeficiency virus (HIV) infection (antibody positive with positive confirmatory molecular test).

2.1.2.2 Patients who have chronic hepatitis B or hepatitis C.

2.1.2.13 Patients with an uncontrolled serious infection.

2.1.2.14 Pregnant or breastfeeding women.

2.1.2.15 Patients with significant medical comorbidities, including uncontrolled hypertension (diastolic blood pressure (BP) greater than 115 mmHg), unstable angina, congestive heart failure (greater than New York Heart Association (NYHA) class II), poorly controlled diabetes, severe chronic pulmonary disease, coronary angioplasty or myocardial infarction within the last 6 months, or uncontrolled atrial or ventricular cardiac arrhythmias.

2.1.2.16 Patients with a history of a psychiatric disorder that may interfere with the understanding and compliance with this protocol and the required follow up.

2.1.2.17 Exclusion at the discretion of the principal investigator (PI) or delegate if participation to the study is deemed too risky (e.g. clinically significant pleural or pericardial effusion or ascites with possibly increased radio-toxicity).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-10-11 (Actual); Primary Completion 2014-11-16 (Actual); Study Completion 2020-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Conlon, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canellos GP, Anderson JR, Propert KJ, Nissen N, Cooper MR, Henderson ES, Green MR, Gottlieb A, Peterson BA. Chemotherapy of advanced Hodgkin's disease with MOPP, ABVD, or MOPP alternating with ABVD. N Engl J Med. 1992 Nov 19;327(21):1478-84. doi: 10.1056/NEJM199211193272102. PMID 1383821
- [Background] Moskowitz CH, Nimer SD, Zelenetz AD, Trippett T, Hedrick EE, Filippa DA, Louie D, Gonzales M, Walits J, Coady-Lyons N, Qin J, Frank R, Bertino JR, Goy A, Noy A, O'Brien JP, Straus D, Portlock CS, Yahalom J. A 2-step comprehensive high-dose chemoradiotherapy second-line program for relapsed and refractory Hodgkin disease: analysis by intent to treat and development of a prognostic model. Blood. 2001 Feb 1;97(3):616-23. doi: 10.1182/blood.v97.3.616. PMID 11157476
- [Background] Josting A, Engert A, Diehl V, Canellos GP. Prognostic factors and treatment outcome in patients with primary progressive and relapsed Hodgkin's disease. Ann Oncol. 2002;13 Suppl 1:112-6. doi: 10.1093/annonc/13.s1.112. No abstract available. PMID 12078891
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-C-0003.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Yttrium-90-labeled Daclizumab + Chemotherapy
Started | 6
Completed | 4
Not Completed | 2
Not completed — mobilization failure | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Yttrium-90-labeled Daclizumab + Chemotherapy
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.05 (8.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity, customized: Mexican, Puerto Rican, Cuban, Central or South Am. | 2
  Ethnicity, customized: Not provided or available | 2
  Ethnicity, customized: Not Hispanic | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of 90Y-daclizumab With Carmustine, Etoposide, Cytarabine, [Ara-C, Cytosine Arabinoside] and Melphalan (BEAM) and Auto Stem Cell Transplant (ASCT): Phase I Portion
Description: The MTD is defined as the dose level below the dose at which 2 out of 2 to 6 patients at a given dose level develop dose limiting toxicity (DLT). A DLT is defined as patients who develop either a Common Terminology Criteria in Adverse Events (CTCAE) v4.0 grade 3 or greater non-hematologic toxicity, with the exception of fatigue, of more than 5 days duration possibly, probably or definitely related to the infusion of 90Y-daclizumab prior to the start of BEAM chemotherapy (Day - 6) will have developed by definition a dose-limiting toxicity (DLT).
Time Frame: Day 100 post autologous stem cell transplant
Population: MTD was not determined due to low enrollment into the study.
Arm/Group | Yttrium-90-labeled Daclizumab + Chemotherapy
Number analyzed (Participants) | 0

2. Primary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: 30 months
Measure: Count of Participants; unit: Participants
Arm/Group | Yttrium-90-labeled Daclizumab + Chemotherapy
Number analyzed (Participants) | 6
Participants | 3

3. Primary Outcome: Number of Participants With A Dose Limiting Toxicity
Description: Patients who develop either a Common Terminology Criteria in Adverse Events (CTCAE) v4.0 grade 3 or greater non-hematologic toxicity, with the exception of fatigue, of more than 5 days duration possibly, probably or definitely related to the infusion of 90Y-daclizumab prior to the start of Carmustine, Etoposide, Cytarabine, [Ara-C, Cytosine Arabinoside] and Melphalan (BEAM) chemotherapy (Day - 6) will have developed by definition a dose-limiting toxicity (DLT).
Time Frame: 30 months
Measure: Count of Participants; unit: Participants
Arm/Group | Yttrium-90-labeled Daclizumab + Chemotherapy
Number analyzed (Participants) | 6
Participants | 0

4. Secondary Outcome: Overall Response Rate
Description: Overall response rate is defined as the number of complete and partial responses in patients with refractory or relapsed Hodgkin's disease. Response is assessed by the Revised Response Criteria for Malignant Lymphoma. Complete response requires all of the following: complete disappearance of all detectable clinical evidence of disease and disease related symptoms if present before therapy. A post treatment residual mass is permitted as long as it is positron emission tomography negative. Partial response requires all of the following: at least a 50% reduction in the sum of the product of the diameters of up to 6 of the largest dominant nodes or nodal masses. These nodes or masses should be selected according to all of the following: they should be clearly measurable in at least two perpendicular dimensions; if possible they should be from disparate regions of the body; and they should include mediastinal and retroperitoneal areas of disease whenever these sites are involved.
Time Frame: Response is evaluated at day 100 post autologous stem cell transplant, then 1-4 times yearly for 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Yttrium-90-labeled Daclizumab + Chemotherapy
Number analyzed (Participants) | 4
Participants
  Complete Response (CR) | 2
  Partial Response (PR) | 2

5. Secondary Outcome: Complete Response Rate
Description: Complete response rate is defined as the time it takes a participant to achieve a complete response. Response is assessed by the Revised Response Criteria for Malignant Lymphoma. Complete response requires all of the following: complete disappearance of all detectable clinical evidence of disease and disease related symptoms if present before therapy. A post treatment residual mass is permitted as long as it is positron emission tomography (PET) negative. If a pretreatment PET scan was negative, all lymph nodes and nodal masses must have regressed on computed tomography (CT) to normal size (<1.5 cm in their greatest transverse diameter for nodes >1.5 cm before therapy); Previously involved nodes that were 1.1 to 1.5 cm in their long axis and more than 1.0 cm in their short axis before treatment must have decreased to <1.0 cm in their short axis after treatment.
Time Frame: 20 months post autologous stem cell transplant
Measure: Median (Full Range); unit: months
Arm/Group | Yttrium-90-labeled Daclizumab + Chemotherapy
Number analyzed (Participants) | 2
months | 7.5 [6 to 9]

6. Secondary Outcome: Disease Free Survival (DFS)
Description: DFS is defined as the amount of time participants remain disease free.
Time Frame: DFS is evaluated at day 100 post autologous stem cell transplant, then 1-4 times yearly for 5 years
Measure: Median (Full Range); unit: months
Arm/Group | Yttrium-90-labeled Daclizumab + Chemotherapy
Number analyzed (Participants) | 4
months | 36 [30 to 42]

7. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the date of registration to the date of death due to any cause or if no death occurs to the last documented information on the patient.
Time Frame: OS is evaluated at day 100 post autologous stem cell transplant, then 1-4 times yearly for 5 years
Measure: Median (Full Range); unit: months
Arm/Group | Yttrium-90-labeled Daclizumab + Chemotherapy
Number analyzed (Participants) | 4
months | 36 [30 to 42]

ADVERSE EVENTS:
Time Frame: 30 months
Arm/Group | Yttrium-90-labeled Daclizumab + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yttrium-90-labeled Daclizumab + Chemotherapy (N=6)
Menopause (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yttrium-90-labeled Daclizumab + Chemotherapy (N=6)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 3 (6)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Infections and infestations - Other, strep mitis bacteremia (Infections and infestations) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (3)
Metabolism and nutrition disorders - Other, Low zinc (Metabolism and nutrition disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nervous system disorders - Other, convulsive syncopal episode (Nervous system disorders) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT01468311/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/11/NCT01468311/ICF_001.pdf